CLINICAL TRIAL: NCT04944342
Title: Thoracal Motion After COVID-19 Disease
Brief Title: Breathing After COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Hilal Hotaman, Assoc Prof, Trakya University
Other Study IDs: 2021/64
Record Dates: First submitted 2021-06-16; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Gait; Covid19; Thorax Anomalies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals who have had COVID-19.: Individuals who have had COVID-19 and who treated by a standart medical treatment at home.
  Interventions: Other: No intervention.
- Individuals who have not a COVID-19 illness history.: Individuals who have not a COVID-19 illness history.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
This research; It will be done to perform thoracic movement analysis of young adult individuals who have survived COVID-19 and to compare them with those without a history of COVID-19.

DETAILED DESCRIPTION:
This research; It will be done to perform thoracic movement analysis of young adult individuals who have survived COVID-19 and to compare them with those without a history of COVID-19.

Individuals' sternal movements using motion analysis sensors; will be recorded in sitting position, standing, and walking. Sternal movement of the person; It will be recorded during relaxed breathing and deep breathing. They will also be asked to walk on the treadmill in such a way as to collect at least 500 steps.

ELIGIBILITY:
Inclusion Criteria:

* to be voluntary.
* have COVID-19 illness history.
* No COVID-19 illness history.
* treated by a standard medical treatment (vitamins, blood thinners, anti-viral drugs)

Exclusion Criteria:

* have another chronic disease such as systemic, orthopedic or neurologic.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals who have a COVID-19 illness history or have no COVID-19 history will be the participants of the study.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Thoracal motion while normal breathing at sitting. | At first day.
  Sensor - based thoracal motion assesment while normal breathing at sitting will be utilized.
Thoracal motion while normal breathing at standing. | At first day.
  Sensor - based thoracal motion assesment while normal breathing at standing will be utilized.
Thoracal motion while deep breathing at sitting. | At first day.
  Sensor - based thoracal motion assesment while normal breathing at sitting will be utilized.
Thoracal motion while deep breathing at standing. | At first day.
  Sensor - based thoracal motion assesment while deep breathing at standing will be utilized.
Thoracal motion at walk. | At first day.
  Sensor - based thoracal motion assesment at walk will be utilized.

IPD SHARING:
Plan to Share IPD: Undecided